CLINICAL TRIAL: NCT05457127
Title: Obstructive Sleep Apnea Treatment in People Aging With Serious Mental Illness
Brief Title: Obstructive Sleep Apnea Treatment in Serious Mental Illness
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ellen Lee, Assistant Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 800600
Record Dates: First submitted 2022-06-22; First posted 2022-07-13 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Schizoaffective Disorder; Schizophrenia; Bipolar Disorder; Obstructive Sleep Apnea of Adult
Keywords: Serious mental illness; aging; positive airway pressure
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Automatic Positive Airway Pressure (APAP) device (Experimental)
  Interventions: Device: Automatic Positive Airway Pressure (APAP)

INTERVENTIONS:
Device: Automatic Positive Airway Pressure (APAP) — If eligible, participants will be given a clinical Automatic Positive Airway Pressure (APAP) device for up to 3 months, while they are waiting for their clinical evaluation from a sleep physician. The APAP device will we will be using is the ResMed Airsense 11 Autoset. APAP is a smart positive airway pressure (PAP) device, where the pressure changes as needed to provide optimal pressure to splint the upper airway. Dr. Lee and Dr. Schmickl will oversee management of the device.
  During the first month of APAP use, individuals will participate in weekly phone calls or in-person visits to ensure optimal adherence and troubleshoot any issues (improper mask fitting, discomfort, etc) that may arise.

SUMMARY:
Serious mental illnesses (SMI) like schizophrenia and bipolar disorder are two of the most disabling and costly chronic illnesses worldwide. A high proportion of adults with schizophrenia and bipolar disorder have sleep disorders, like obstructive sleep apnea (OSA), but tend to be underdiagnosed and undertreated compared to the general population. This study aims to examine feasibility, acceptance, and impact of OSA treatment and how it affects cognitive function in people with SMI.

DETAILED DESCRIPTION:
Sleep disturbances are central to many psychiatric disorders, including schizophrenia and bipolar disorder, with clear implications for cognition, brain health, physical health and aging. Obstructive sleep apnea (OSA) is typically underdiagnosed and undertreated due to impairment from psychiatric symptoms, limited resources, and stigma. In turn, consequences of untreated OSA in SMI are dire: in particular, worsening cardiometabolic health, cognitive decline, and death. Few studies have examined the impact of treatments for obstructive sleep apnea on cognitive problems in a high-risk group, such as older adults with SMI. The goals of the proposed study are to assess the acceptance and effectiveness of positive airway pressure (PAP) treatment for OSA, and its impact on cognitive and cardiometabolic outcomes as well as biological processes over a 3-month period. In order to determine eligibility, participants will be asked to complete a diagnostic test either at home or overnight in-lab. If diagnosed with sleep apnea, the participant will be offered a 3-month treatment with an automatic PAP. In addition, eligible participants will complete weekly check-ins with study staff and a series of detailed interviews, physical and neuropsychological tests, instrumental and clinical assessments, and blood draws every month for a total of 3 months.

ELIGIBILITY:
Inclusion Criteria:

Control participants:

* lifetime absence of major psychiatric illness
* 40 to 70 years old
* be at risk for or have a diagnosis of obstructive sleep apnea

For participants with serious mental illness:

* diagnosis of schizophrenia, schizoaffective disorder, or bipolar disorder
* must not be conservatized
* 40 - 70 years old
* be at risk or have a diagnosis of obstructive sleep apnea.

Exclusion Criteria:

* DSM-IV-TR diagnosis of active alcohol or other substance abuse or dependence in the 3 months preceding enrollment. This will be self-report.
* Diagnosis of dementia, mental retardation, or other neurological or medical conditions known to affect neurophysiologic or neurocognitive functioning, or autoimmune disease
* Other major DSM-IV-TR Axis I Disorder
* Medical problems that interfere with a participant's ability to complete the assessments
* Plans to move out of the San Diego county area within the following 6 months
* Diagnosis of OSA and currently receiving APAP, CPAP, or any treatment from a physician.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Acceptance of PAP trial | 3 months
  Acceptance of PAP trial (based on post-adherence program survey taken after the completion of the 4 sessions.) Acceptability will be rated by % individuals who rate high level of satisfaction with the intervention.
OSA self-efficacy using the SEMSA | 3 months
  OSA self-efficacy will be assessed using the Self-Efficacy Measure for Sleep Apnea (SEMSA). The SEMSA is a 26-item, self-administered questionnaire. The SEMSA has 3 categories: perceived risk, outcome expectancies, and treatment self-efficacy. In the perceived risk category, individuals answer questions about their perceived vulnerability to health risks. In the outcome expectancies, individuals answer questions regarding the potential behavior to reduce those risks, and in the treatment self-efficacy, the participant rates the level of validity of the statements on a 4-point scale regarding their perceived ability to perform behavior. Each of the 3 categories has a 4-point ordinal scale (1= irrelevant, 4 = extremely relevant) ranging from very low to very high. The mean of the 3 subscales are calculated. Higher scores indicate greater perceived self-efficacy, perceived response efficacy, and higher perceived susceptibility.
PAP usage | 3 months
  PAP usage will be assessed using mean hours/night - which will be obtained from the PAP machine data.
Cognitive Functioning | 3 months
  Cognitive functioning will be measured with the MATRICS Cognitive Consensus Battery (MCCB).159 The MCCB assesses six cognitive domains (attention/vigilance**, verbal learning/memory**, processing speed, working memory, auditory learning/memory, and reasoning), and has excellent test-retest reliability (ICC = 0.88) with minimal practice effects.159, 160 Executive functioning is the one cognitive domain that is less ideally covered within the MCCB. The closest MCCB domain, reasoning, is measured by a single timed-mazes task that can be readily affected by non-executive functions. We use subtests from the Delis-Kaplan Executive Functioning System (D-KEFS) battery161 [Color Word Interference, Letter Number Sequencing, and phonemic (FAS) and semantic (Animals) fluency] to assess Executive Functioning*. We have successfully employed these measures as a supplement to the MCCB in multiple prior studies in PwS.
Monitoring Slow Wave Sleep and Sleep Spindle Density | 3 months
  Slow wave sleep -based on proportion/duration of Slow wave activity on overnight sleep EEG recordings. Sleep Spindle density - based on sleep spindle density measured during non-REM sleep on overnight sleep EEG recordings

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, La Jolla, California, United States